CLINICAL TRIAL: NCT02640222
Title: APIXABAN in the Prevention of Stroke and Systemic Embolism in Patients With Atrial Fibrillation in Real-Life Setting in France SNIIRAM Study
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-285
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Anticoagulation
MeSH Terms: interventions — acarboxyprothrombin; apixaban; Dabigatran; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- AC-naive treated with VKA: AC-naive treated with VKA
  Interventions: Drug: VKA
- AC-naive treated with apixaban: AC-naive treated with apixaban
  Interventions: Drug: Apixaban
- AC-naive treated with dabigatran: AC-naive treated with dabigatran
  Interventions: Drug: dabigatran
- AC-naive treated with rivaroxaban: AC-naive treated with rivaroxaban
  Interventions: Drug: rivaroxaban
- AC-experienced treated with VKA: AC-experienced treated with VKA
  Interventions: Drug: VKA
- AC-experienced treated with apixaban: AC-experienced treated with apixaban
  Interventions: Drug: Apixaban
- AC-experienced treated with dabigatran: AC-experienced treated with dabigatran
  Interventions: Drug: dabigatran
- AC-experienced treated with rivaroxaban: AC-experienced treated with rivaroxaban
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: VKA
  Other Names: Vitamin K antagonist
  Groups: AC-experienced treated with VKA; AC-naive treated with VKA
Drug: Apixaban
  Groups: AC-experienced treated with apixaban; AC-naive treated with apixaban
Drug: dabigatran
  Groups: AC-experienced treated with dabigatran; AC-naive treated with dabigatran
Drug: rivaroxaban
  Groups: AC-experienced treated with rivaroxaban; AC-naive treated with rivaroxaban

SUMMARY:
The purpose of this study is to evaluate the APIXABAN use in the Prevention of Stroke and Systemic Embolism in Patients with Atrial Fibrillation in Real-Life Setting in France, data from SNIIRAM (French data base).

ELIGIBILITY:
Inclusion Criteria:

* Patient meeting inclusion criteria of the French Système national d'information inter-régimes de l'assurance maladie (SNIIR-AM)/Programme de médicalisation des systèmes d'information (PMSI) claim databases (Patient insured by the French national health insurance general scheme stricto sensu (apart from local mutualist sections)
* Patients with at least one reimbursement of AC treatment (acenocoumarol, warfarine and fluidione for VKA treatments, apixaban, dabigatran or rivaroxaban for New oral anticoagulants (NOACs)) treatments during the inclusion period
* Patients initiated with a new AC treatment during the inclusion period, either AC naive or not
* Patients aged 18 or older at their first anticoagulant initiation during the inclusion period
* Patient diagnosed with non-valvular Atrial fibrillation (AF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AC-naive and AC-experienced patients diagnosed with non-valvular AF, initiated with either apixaban, dabigatran, rivaroxaban or VKAs
Sampling Method: Non-Probability Sample
Enrollment: 321501 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of first event of stroke and/or systemic embolism over the period of AC exposure | Approximately 2 years
  Estimation by AC treatment and for both populations (AC-naive and AC-experienced patients) of Incidence rate (95%CI) of first event of stroke and/or systemic embolism (effectiveness) and of first event of major bleeding (safety) over the period of AC ex
Time-to-first occurrence of stroke or systemic embolism will be estimated and plotted using Kaplan-Meier product limit estimator | Approximately 2 years
  Estimation by AC treatment and for both populations (AC-naive and AC-experienced patients) of Time-to-first occurrence of stroke and/or systemic embolism (effectiveness) and of major bleedings (safety) using Kaplan-Meier product limit estimator (95%CI)

SECONDARY OUTCOMES:
Incidence rates for composite morbidity criterion and all-cause death over the period of AC exposure will be estimated by AC treatment | Approximately 2 years
  * Risk of occurrence of a composite morbidity criterion: number of patients presenting at least 1 event during the exposure period, incidence rate, median time to occurrence of event in each subcohort, composite morbidity criterion being defined by stroke, systemic embolism or major bleeding, whichever occurs first.
  * Risk of all-cause mortality: number of deaths during exposure period to studied AC treatment, incidence rate, median survival time
Time-to-event for composite morbidity criterion and all-cause death using Kaplan-Meier product limit estimator (95%CI) | Approximately 2 years
Major characteristics of patients will be described by AC treatments | Approximately 2 years
  Major characteristics of patients and comorbidities were:
  * proportion of AC-naive patients by AC treatment
  * In each subcohort:
    * Sociodemographic characteristics: median age, sex ratio, region of residence, CMU-C (Universal Health Coverage Complementary) beneficiary,
    * NVAF characteristics : time since NVAF diagnosis,
    * ALD status distribution (ALD Type, ICD-10 code for diagnosis),
    * Past hospital stay : number and total length of hospital stays
    * Previous exposure to AC treatment (class, molecule) over the 3 previous years, for AC-experienced patients.
    * Thromboembolism risk factors: CHADS2 mean score, CHA2DS2 VASc mean score, and distribution according to the scores.
    * Bleeding risk factors: modified HASBLED mean score and distribution according to the scores
    * Charlson mean score and distribution according to the scores
Treatment patterns at AC initiation, over time and concomitant treatment will be tabulated by AC treatment | Approximately 2 years
  Treatment patterns at AC initiation: Type of the prescriber initiating the AC treatment (general practitioners, office-based cardiologists, hospital-based physicians and others), prescribed dosages, duration of initial prescription, co prescription (others AC, antiplatelet agents, NSAIDs, SRIs, strong inhibitors of both CYP3A4, anticonvulsivant strong inducer of hepatic enzymes, rifampicine, antiarrhythmic drugs)
Time-to-discontinuation will be estimated and plotted using Kaplan-Meier product limit estimator | Approximately 2 years
  Time-to-discontinuation will be estimated and plotted using Kaplan-Meier product limit estimator based on Adherence to treatment: mean Medication Possession Ratio (MPR), Persistence: number for AC treatment discontinuation, median time to discontinuation
The healthcare resources utilization will be described by AC treatment | Approximately 2 years
  The healthcare resources utilization will be described by AC treatment based on number of medical visits, number of nurse acts, per category of act, number of drugs packages per therapeutic classes, number of biology and tests, per type of act, number of other explorations, number of hospital stays, number of sick leaves
Comparisons of major characteristics of patients between apixaban and each of the other AC treatments | Approximately 2 years
  Comparisons of major characteristics of patients between apixaban and each of the other AC treatments will be performed using:
  * An analysis adjusted for confounding factors in order to verify adjustment quality and using:
    * the Wald test from a logistic regression model for binary and other qualitative variables
    * the F- test from a covariance analysis for quantitative variables
  * An analysis after matching for confounding factors in order to verify matching quality and using:
    * the Cochran-Mantel-Haenzel test for qualitative variables
    * the F-test from a covariance analysis for quantitative variables
Comparison of incidence rates of each studied event (stroke or systemic thromboembolic event, major bleeding, all-cause death) between apixaban and each of the other usual AC treatments | Approximately 2 years
Comparative time-to-event analyses for each studied event between apixaban and each of the other usual AC treatments | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Rueil-Malmaison, France

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm